CLINICAL TRIAL: NCT05883436
Title: A Prospective, Multi-Center Investigation of the DEXA- C Anterior Cervical Interbody System
Brief Title: Investigation of DEXA-C Anterior Cervical Interbody System
Acronym: DEXA-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aurora Spine and Pain (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 01-AUR-DEXA-23
Record Dates: First submitted 2023-04-04; First posted 2023-06-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Degenerative Disc Disease
Keywords: fusion; subsidence
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: The Dexa-C Study will be conducted at up to 10 investigative sites in the United States. It is anticipated that at least 40 single level subjects and at least 40 multiple level subjects will be enrolled into the Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm Observational (Other): Cervical Interbody Cage
  Interventions: Device: DEXA-C Cervical Interbody System

INTERVENTIONS:
Device: DEXA-C Cervical Interbody System — The Dexa-C Cervical Interbody System is intended for use on patients who require anterior cervical discectomy and fusion surgery. The system implants an interbody spacer(s) into the cervical intervertebral body space(s) to stabilize and fuse the level(s). Allograft will be used in the spacer and the spinal segment(s) are fixed with an anterior cervical plate

SUMMARY:
FDA Cleared interbody product for the cervical spine, designed to match a patients DEXA scan for increase in fusion rate.

DETAILED DESCRIPTION:
The DEXA-C Cervical Interbody System is indicated for anterior cervical interbody fusion procedures in skeletally mature patients with degenerative disc disease (DDD) of the cervical spine with accompanying radicular symptoms at one or two contiguous levels from C2-T1. Device system is designed for use with supplemental fixation and autograft and/or allogenic bone graft composed of cancellous, cortical, and/or cortico-cancellous bone to facilitate fusion and is to be implanted via an open, anterior approach. The Dexa-C clinical study will collect data on those patients who have been treated with Dexa-C Anterior Cervical Interbody System to allow for a better understanding of outcomes associated with it.

ELIGIBILITY:
Inclusion Criteria:

1. Must already be scheduled or planned for anterior cervical discectomy and fusion using the Dexa-C Anterior Interbody System C3-7 with supplemental fixation and/or allogenic bone graft composed of cancellous, cortical, and/or cortico-cancellous bone meeting on-label criteria.
2. Radicular signs and symptoms in one or both arms (i.e., pain, paresthesia or paresis in a specific nerve root distribution).
3. Diagnosis of cervical radiculopathy at one or two contiguous levels from C3-7 requiring open anterior cervical fusion and discectomy.
4. Diagnosis of degenerative disc disease by radiographic evidence of cervical disc herniation and/or osteophytes accompanying clinical symptoms.
5. At least 6 weeks prior conservative treatment (i.e. physical therapy, pain medication).

Exclusion Criteria:

1. History of cervical spine surgery less than 12 months prior to surgery.
2. Diagnosis of severe spondylosis.
3. Patients requiring posterior cervical surgery, anterior cervical corpectomy, or revision surgery.
4. Any member of a vulnerable population (ie. minors, adults who lack the ability to consent, pregnant women, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-22 (Estimated)

PRIMARY OUTCOMES:
Fusion Assesment | 12 months
  The primary outcomes of interest for this study will be fusion assessment at 3 months, 6 months and 12 months post-surgery.
  Fusion assessment from Static and Dynamic X-Ray (AP/LAT/Flex/Ex) using the following criteria:
  Bridging bone inside or outside of graft No lucencies at the graft-vertebral body junction Motion < 1mm

SECONDARY OUTCOMES:
Subsidence | 12 months
  Secondary outcome measures will include subsidence. Patient reported outcomes (Neck Disability Index on a 0-50 scale (NDI) and Visual Analog Scale for Pain (VAS) on a 0-10 scale will be collected at follow up visits and assessed compared to baseline.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCI Center for Clinical Research, Orange, California
  - Orthopaedic Institute of Western KY, Paducah, Kentucky
  - Koga Neurosurgery, Covington, Louisiana
  - Optima Orthopedics, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No